CLINICAL TRIAL: NCT04358328
Title: Effect of CGA for Frail Elderly Patients Operated for Colorectal Cancer - The CRC Frailty-study Can Preoperative Comprehensive Geriatric Assessment and Care in Addition to Standard ERAS Protocol Reduce Mortality After Colorectal Surgery for Carcinoma in the Frail Elderly?
Brief Title: Effect of CGA for Frail Elderly Patients Operated for Colorectal Cancer - The CRC Frailty-study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Mattias Prytz, Senior Consultant surgeon, MD, PhD. Head of the Colorectal department, Department of Surgery, NU-Hospital Organization, Sweden, NU-Hospital Organization, Sweden
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Frailty-studien
Record Dates: First submitted 2020-04-02; First posted 2020-04-24 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Colorectal Neoplasms; Frailty; CGA
Keywords: Frailty; Elderly; Colorectal cancer; Comprehensive Geriatric Assessment
MeSH Terms: conditions — Colorectal Neoplasms; Frailty | interventions — Geriatric Assessment; Standard of Care

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into two parallel groups. This will result in two equally sized groups which will be stratified for the planned surgical procedure (colon- or rectal surgery), gender and age. One group will be randomized to preoperative geriatric-, nursing-, physiotherapist-, and dietician assessments followed by appropriate interventions (CGA and care). The other group will be randomized to conventional preoperative assessments by anaesthesiologist and standard ERAS care. The study population is constituted of all patients in the participating hospitals with a newly diagnosed colorectal cancer available for colorectal cancer surgery with curative intent and who fulfil the inclusion criteria and no exclusion criteria.
Who Masked: Outcomes Assessor
Masking Description: It will not be possible to mask for either patients nor participating health care professionals if patients are enrolled in the control- or intervention group. Hence, the study will not be blinded. When the final data analysis is performed the person performing the analysis will not be aware of which group each patient was a part of.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The patients in the intervention arm will receive the same care and treatment as is provided to all patients in the clinical setting, including the ERAS-concept. In addition to this they will be individually assessed by a physician with geriatric profile, dietician, physiotherapist and nurse and thereafter undergo appropriate interventions (CGA and care). The intervention team will have weekly meetings regarding the patients included in the study to evaluate how long the intervention should continue before surgery, a maximum time of eight weeks will be allowed for the intervention.
  Interventions: Other: Comprehensive geriatric assessment (CGA) and care
- Control group (Active Comparator): The patients in the control group will standard care and treatment which include assessment of surgeons, anaesthesiologists and, if needed, other specialized physicians. They will be treated according to the ERAS-concept in the pre- peri- and post operative phase.
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Comprehensive geriatric assessment (CGA) and care — Comprehensive geriatric assessment and care including geriatric-, nursing-, physiotherapist-, and dietician assessments followed by appropriate interventions.
  Arms: Intervention group
Other: Standard care — Standard pre-, peri- and post operative care.
  Arms: Control group

SUMMARY:
This multicentre randomized controlled trial aims to investigate whether an individualized comprehensive geriatric assessment (CGA) and care will improve postoperative results in frail elderly patients undergoing surgery for colorectal cancer. The study will take place in departments applying the ERAS-concept which is considered gold standard in colorectal surgery.

DETAILED DESCRIPTION:
Colorectal cancer is the third most common cancer form in Sweden with an incidence of approximately 6000 new cases annually. It affects mainly elderly people; 65 % of patients diagnosed with colon- or rectal cancer are older than 65 years, and more than half are 70 years of age or older when diagnosed. Surgery is the treatment of choice for colon and rectal cancer if cure is to be achieved, sometimes in combination with radio- and/or chemotherapy. With increasing age many patients acquire other medical conditions which in turn can affect the patient's general status and thus impair their chances to recover from cancer treatment.

Age is a well-known risk factor for post-operative complications. Furthermore, it has been established that assessing frailty in elderly patients is a more precise way of detecting patients with increased vulnerability. In recent years increasing research has focused on frailty in regards of different medical conditions and treatments. A large amount of studies has also been conducted on the concept of frailty and surgery, and there is solid knowledge of the impact of frailty on outcome after surgery. It is also known that elderly frail patients suffers a higher risk of severe post-operative complications and morbidity compared to elderly non frail patients in the terms of elective surgery for colon- and rectal cancer.

Several different tools for determining and measuring frailty has been developed and studied. A commonly used definition is the accumulation of deficits model, which adds together a person's different diseases and disabilities. A widely used instrument based on this concept is the Canadian Study of Health and Aging (CSHA) Clinical Frailty Scale (CFS-9). It utilises a 9-point instrument to assess frailty. A score of 5 or more defines frailty, and the higher the score the more severe the degree of frailty. The instrument has been extensively studied and validated and is highly correlated to the degree of frailty as measured with much more extensive frailty tools. The instrument is easy to use and not very time-consuming which makes it practical to use in everyday clinical practice; therefore rendering it relevant to use in clinical studies.

As stated, there are evidence that the group of frail elderly patients have inferior results after colorectal surgery, compared to elderly non-frail patients. Comprehensive geriatric assessment (CGA) and care is a well-established and effective way of providing health care. It has been proven to be beneficial in terms of outcome after hospitalization for the group of frail elderly in various other settings. A multicentre randomized controlled trial conducted in Norway evaluated preoperative geriatric assessment prior to surgery for colorectal cancer in frail patients ≥ 65 years of age. The patients in the intervention group were assessed by a medical doctor specializing in geriatric medicine who gave individual advice regarding medical changes, exercise, nutrition etc. The median time of intervention before surgery was six days. The study could not show any significant differences in post-operative complications. Except having a brief time span for the intervention, the study was smaller than the initial estimation, with a total of 116 included patients. Another randomized controlled study has been conducted regarding prehabilitation prior to surgery for colorectal cancer in frail patients, analysing 30-day complications. The prehabilitation in this study consisted of exercise, nutritional and psychological interventions four weeks prior to surgery, and could not establish any differences in 30-day complications rates compared to a group that received rehabilitation four weeks after surgery. Further, there is an ongoing randomized controlled international study aiming to evaluate the impact of multimodal prehabilitation - in terms of exercise, nutritional and psychological interventions prior to colorectal surgery in adults, not specifically frail patients. There is also an ongoing randomized controlled study - the GERICO study - on frail elderly patients receiving chemotherapy for colorectal cancer with the aim to see if geriatric intervention affects outcome.

Intervention studies using CGA and care as an intervention to improve outcome for frail elderly patients has been conducted in terms om hip fracture and abdominal surgery, so far with mixed results. A systematic review of these studies from 2017 concluded that there is a need of a larger randomized multicentre study to evaluate the possible advantage of such an intervention for frail elderly patients prior to surgery.

ELIGIBILITY:
Inclusion Criteria:

* Potentially curable colorectal cancer (according to cTNM)
* ≥ 70 years old
* Frailty (CFS-9 v2.0 score 4-8)

Exclusion Criteria:

* Palliative situation
* Unable to understand study information
* Acute surgery
* Terminally ill patient (CFS-9 9)
* Less than 6 months expected survival
* Not willing to participate

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | 90 days
  All cause mortality

SECONDARY OUTCOMES:
Hospital stay | 3 months
  Length of hospital stay and total number of hospital days within 3 months after discharge
Discharge destination | 2 months
  Home or nursing facility, use of home help services. Information regarding where the patient was discharged after the hospital care will be gathered from the medical records. It will be noted if the patient was discharged to: own housing without home help services or home healthcare, own housing with assistance of home help services and/or home healthcare or to a nursing facility.
Readmission | 30 days
  30 days readmission rates
Acitivities of Daily Living (ADL) | 2 months
  ADL performance at follow up in comparison to baseline. ADL performance will be assessed using the ADL Staircase. This instrument evaluates a person's independence regarding nine functions: bathing, dressing, toileting, transferring, feeding, cooking, shopping, cleaning, and transportation. The results gives a score of 0-9 where 9 indicates complete dependence regarding all functions and 0 indicates full function.
Safe medication assessment | 2 months
  Medication assessment at follow-up, by the instrument Safe medication assessment (SMA) and via clincial evalutation.
Clinical Frailty Scale-9 (CFS-9) | 2 months
  CFS-9 score at follow up.
  The CFS-9 scale is a validating scoring system for detecting frailty in elderly. The scale reaches from 0-9, patients reaching a score of 5-8 are considered to be frail. A higher number indicates increased frailty.
Postoperative complications | 2 months
  According to the Clavien-Dindo scale. The Clavien-Dindo scale is a well-recognized tool for grading post-operative complications. The scale reaches from 1-5, where 1 is a minor complication and 5 is a deadly complication.
Quality of Life (QoL) | 12 months
  Health related QoL at follow up, measured using the "EQ-5D-5L"-form. The form evaluates the patients self-experienced degree of mobility, self-care, usual activities, pain/discomfort and anxiety and depression. The scoring results in an index value which can be compared to a standard value of the general population in a region/country.
Health economical calculations | 1 year
  Including cost-effectiveness based on costs of hospital care, primary care and municipal care; mortality, and quality of life (QoL).
Mortality | 1 years
  All cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Mattias Prytz, MD, PhD, Principal Investigator — Department of Surgery, NU-Hospital Organization
Locations (2):
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg, Västra Götalandsregionen
  - Department of Surgery, NU-Hospital/NÄL, Trollhättan, Västra Götalandsregionen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Okabe H, Ohsaki T, Ogawa K, Ozaki N, Hayashi H, Akahoshi S, Ikuta Y, Ogata K, Baba H, Takamori H. Frailty predicts severe postoperative complications after elective colorectal surgery. Am J Surg. 2019 Apr;217(4):677-681. doi: 10.1016/j.amjsurg.2018.07.009. Epub 2018 Nov 23. PMID 30473227
- [Background] Ommundsen N, Wyller TB, Nesbakken A, Bakka AO, Jordhoy MS, Skovlund E, Rostoft S. Preoperative geriatric assessment and tailored interventions in frail older patients with colorectal cancer: a randomized controlled trial. Colorectal Dis. 2018 Jan;20(1):16-25. doi: 10.1111/codi.13785. PMID 28649755
- [Background] Ommundsen N, Wyller TB, Nesbakken A, Jordhoy MS, Bakka A, Skovlund E, Rostoft S. Frailty is an independent predictor of survival in older patients with colorectal cancer. Oncologist. 2014 Dec;19(12):1268-75. doi: 10.1634/theoncologist.2014-0237. Epub 2014 Oct 29. PMID 25355846
- [Background] Tan KY, Kawamura YJ, Tokomitsu A, Tang T. Assessment for frailty is useful for predicting morbidity in elderly patients undergoing colorectal cancer resection whose comorbidities are already optimized. Am J Surg. 2012 Aug;204(2):139-43. doi: 10.1016/j.amjsurg.2011.08.012. Epub 2011 Dec 16. PMID 22178483
- [Background] Rockwood K, Song X, MacKnight C, Bergman H, Hogan DB, McDowell I, Mitnitski A. A global clinical measure of fitness and frailty in elderly people. CMAJ. 2005 Aug 30;173(5):489-95. doi: 10.1503/cmaj.050051. PMID 16129869
- [Background] Reisinger KW, van Vugt JL, Tegels JJ, Snijders C, Hulsewe KW, Hoofwijk AG, Stoot JH, Von Meyenfeldt MF, Beets GL, Derikx JP, Poeze M. Functional compromise reflected by sarcopenia, frailty, and nutritional depletion predicts adverse postoperative outcome after colorectal cancer surgery. Ann Surg. 2015 Feb;261(2):345-52. doi: 10.1097/SLA.0000000000000628. PMID 24651133
- [Background] Pilotto A, Cella A, Pilotto A, Daragjati J, Veronese N, Musacchio C, Mello AM, Logroscino G, Padovani A, Prete C, Panza F. Three Decades of Comprehensive Geriatric Assessment: Evidence Coming From Different Healthcare Settings and Specific Clinical Conditions. J Am Med Dir Assoc. 2017 Feb 1;18(2):192.e1-192.e11. doi: 10.1016/j.jamda.2016.11.004. Epub 2016 Dec 31. PMID 28049616
- [Background] Indrakusuma R, Dunker MS, Peetoom JJ, Schreurs WH. Evaluation of preoperative geriatric assessment of elderly patients with colorectal carcinoma. A retrospective study. Eur J Surg Oncol. 2015 Jan;41(1):21-7. doi: 10.1016/j.ejso.2014.09.005. Epub 2014 Sep 18. PMID 25267000
- [Derived] Normann M, Ekerstad N, Angenete E, Prytz M. Effect of comprehensive geriatric assessment for frail elderly patients operated for colorectal cancer-the colorectal cancer frailty study: study protocol for a randomized, controlled, multicentre trial. Trials. 2022 Nov 17;23(1):948. doi: 10.1186/s13063-022-06883-9. PMID 36397083